CLINICAL TRIAL: NCT06514989
Title: Efficacy of Low-residue Full Nutritive Formula Powder in Bowel Preparation for Colonoscopy: a Multicenter Non-inferiority Randomized Controlled Study
Brief Title: Efficacy of Low-residue Full Nutritive Formula Powder in Bowel Preparation for Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of the Department of Gastroenterology, the First Affiliated Hospital of Naval Medical University, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: FNFP2024
Record Dates: First submitted 2024-07-18; First posted 2024-07-23 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Bowel Preparation for Colonoscopy
Keywords: Bowel preparation, Low-residue diet, colonoscopy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-residue nutrition formula podwer combined with 2 liters of polyethylene glycol (Experimental)
  Interventions: Dietary Supplement: Low-residue full nutrition formula podwer
- Self-prepared low-residue diet combined with 3 liters of polyethylene glycol (Active Comparator)
  Interventions: Dietary Supplement: Self-prepared low-residue diet

INTERVENTIONS:
Dietary Supplement: Low-residue full nutrition formula podwer — The day before the colonoscopy, subjects were given a low-residue full nutrition formula podwer instead of a traditional self-prepared low-residue diet. Subjects were given 6 packs (60g/pack) pre-packaged FNFP and asked to use the FNFP according to individual needs. The 2 liters of polyethylene glycol solution is taken in split dosing, with 1 liter taken at 8pm the day before the colonoscopy and 1 liter taken 3-5 hours before the colonoscopy.
  Arms: Low-residue nutrition formula podwer combined with 2 liters of polyethylene glycol
Dietary Supplement: Self-prepared low-residue diet — Subjects in the self-prepared Low-residue diet group were instructed to follow and prepare an Low-residue diet in the day prior to colonoscopy. The 3 liters of polyethylene glycol solution is taken in split dosing, with 1 liter taken at 8pm the day before the colonoscopy and 2 liter taken 4-6 hours before the colonoscopy.
  Arms: Self-prepared low-residue diet combined with 3 liters of polyethylene glycol

SUMMARY:
Previously, our team compared the effects of a low-residue full nutrition formula podwer (FNFP) combined with 3 liters of polyethylene glycol(PEG) solution and the self-prepared low-residue diet combined with 3 liters of PEG solution on the quality of bowel preparation for colonoscopy, and the results showed that the adequate bowel preparation rate was significantly improved in low-residue full nutrition formula podwer group. However, there are still a considerable number of patients in the process of taking 3L PEG appeared bloating, abdominal pain, nausea, vomiting and other adverse reactions, indicating some subjects can not tolerate the dosage of 3L PEG. In order to reduce adverse reactions and provide more options for people with low PEG tolerance, this study intends to compare the effects of low-residue FNFP combined with 2L PEG and self-provided low-residue diet combined with 3L PEG on the quality bowel preparation, colonoscopy lesions detection, adverse reactions, and tolerance, compliance and satisfaction of subjects.

ELIGIBILITY:
Inclusion Criteria:

* adult subjects between the ages of 18 and 75 who were scheduled for screening, monitoring, and diagnostic colonoscopy.

Exclusion Criteria:

* severe heart, brain, lung, kidney complications or a history of acute myocardial infarction within six months.
* a history of abdominal or pelvic surgery, BMI > 28 or BMI < 18.5, inflammatory bowel disease, constipation (less than 3 bowel movements in the past week, with strenuous bowel movements, hard stool, small volume), or intestinal obstruction.
* imaging and laboratory tests are highly suspicious of colorectal cancer or warning signs and symptoms of colorectal cancer: blood in the stool, black stool, unexplained anemia and significant weight loss, abdominal mass, and positive digital rectal examination.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 757 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Adequate bowel preparation rate | Two months
  Defined as score ≥ 2 for all colon segment (right-side colon, transverse colon, and left-side colon) according to the Boston Bowel Preparation Scale

SECONDARY OUTCOMES:
Excellent bowel preparation rate | Two months
BBPS score (including total score, left colon, transverse colon, and right colon) | Two months
Aronchick Scale score | Two months
Bowel preparation completion rate | Two weeks
  PEG intake is more than 90% of the requirement
Subject satisfaction rate | Two weeks
Colonoscopist satisfaction rate | Two weeks
Adenoma detection rate | Four weeks
Polyp detection rate | Two weeks
Compliance with FNFP | Two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhaoshen, PhD, Study Chair — Department of Gastroenterology, Changhai Hospital, Navy Medical University
Locations (27):
- China (27):
  - Lu'an People's Hospital, Lu'an, Anhui
  - PLA 909 Hospital, Quanzhou, Fujian
  - PLA 909 Hospital, Zhangzhou, Fujian
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Hebei North University, Zhangjiakou, Hebei
  - Jiangsu Provincial Hospital of Traditional Chinese Medicine, Nanjin, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing Gulou Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - Jiangsu Subei People's Hospital, Yangzhou, Jiangsu
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - the central hospital of Dalian, Dalian, Liaoning
  - Northern Theater General Hospital, Shenyang, Liaoning
  - Shengli Oilfield Central Hospital, Dongying, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Changhai Hospital, Naval Medical University, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Ankang Central Hospital, Ankang, Shanxi
  - Yibin Second People's Hospital, Yibin, Sichuan
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - East China Hospital, Fudan University, Shanghai
  - Shanghai Seventh People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No